CLINICAL TRIAL: NCT07058402
Title: A Multicenter, Randomized Controlled Trial Comparing the Retrograde Intrarenal Surgery With a Tip-Flexible Suction Access Sheath to the Standard Percutaneous Nephrolithotomy for the Treatment of 2-3 cm Unilateral Renal Stones
Brief Title: RIRS With Flex Suction Sheath vs. PCNL for 2-3 cm Renal Stones
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Zhejiang Provincial People's Hospital (Other); Affiliated Hospital of Jiaxing University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20250408
Record Dates: First submitted 2025-05-28; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-04

CONDITIONS: Nephrolithiasis
Keywords: Renal Calculi; Percutaneous Nephrolithotomy; PCNL; Retrograde Intrarenal Surgery; RIRS; Flexible Suction Access Sheath
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrograde Intrarenal Surgery (RIRS) with Tip-Flexible Suction Access Sheath (Experimental): Participants in this group will undergo retrograde intrarenal surgery (RIRS) using a tip-flexible suction access sheath for the treatment of 2-3 cm unilateral renal stones.
  Interventions: Procedure: Retrograde Intrarenal Surgery (RIRS) with Tip-Flexible Suction Access Sheath
- Standard Percutaneous Nephrolithotomy (PCNL) (Experimental): Participants in this group will undergo standard percutaneous nephrolithotomy (PCNL) for the treatment of 2-3 cm unilateral renal stones.
  Interventions: Procedure: Standard Percutaneous Nephrolithotomy (PCNL)

INTERVENTIONS:
Procedure: Retrograde Intrarenal Surgery (RIRS) with Tip-Flexible Suction Access Sheath — Participants undergo retrograde intrarenal surgery (RIRS) using a tip-flexible suction access sheath. The procedure involves the insertion of a flexible ureteroscope through the urethra and ureter into the kidney. A novel access sheath with tip-flexible and suction capabilities is used to facilitate stone fragmentation and removal. The goal is to improve stone clearance and reduce intrarenal pressure during the procedure.
  Arms: Retrograde Intrarenal Surgery (RIRS) with Tip-Flexible Suction Access Sheath
Procedure: Standard Percutaneous Nephrolithotomy (PCNL) — Participants undergo standard percutaneous nephrolithotomy (PCNL). The procedure involves creating a percutaneous tract into the renal collecting system under imaging guidance, followed by nephroscope insertion to fragment and extract 2-3 cm renal stones. This represents the current standard of care for large renal calculi.
  Other Names: RIRS with Tip-Flexible Suction Access Sheath
  Arms: Standard Percutaneous Nephrolithotomy (PCNL)

SUMMARY:
This is a multicenter, randomized controlled trial comparing retrograde intrarenal surgery (RIRS) using a tip-flexible suction access sheath with standard percutaneous nephrolithotomy (PCNL) for the treatment of 2-3 cm unilateral renal stones. The aim is to evaluate the clinical efficacy and safety of the novel suction sheath-assisted RIRS compared to standard PCNL in terms of stone-free rate and postoperative complications. A total of 308 patients will be enrolled across four centers in China.

DETAILED DESCRIPTION:
Kidney stones (renal calculi) are a common urological condition that can lead to pain, infection, and renal dysfunction. For renal stones measuring 2-3 cm, both retrograde intrarenal surgery (RIRS) and percutaneous nephrolithotomy (PCNL) are recognized treatment options. Traditional RIRS is less invasive but may be associated with lower stone-free rates for larger stones. A newly developed tip-flexible suction access sheath (TFS-UAS) allows improved access to renal calyces, reduces intrarenal pressure, and enables efficient stone fragment evacuation through continuous suction.

This study is a prospective, multicenter, randomized controlled trial designed to compare the effectiveness and safety of RIRS using the TFS-UAS versus standard PCNL in patients with unilateral renal stones measuring 2-3 cm. A total of 308 patients aged 18-80 years will be enrolled from four tertiary hospitals in China. Eligible participants will be randomized into two groups to receive either TFS-UAS-assisted RIRS or standard PCNL. The primary endpoint is the stone-free rate (SFR) at 3 months, assessed by CT scan. Secondary outcomes include postoperative infection rates, changes in hemoglobin and procalcitonin levels, hospital stay duration, and pain scores.

This study aims to provide high-quality evidence to guide surgical decision-making in the management of medium-sized kidney stones and to evaluate the potential advantages of the new suction-assisted sheath in minimally invasive endourology.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years
2. American Society of Anesthesiologists (ASA) physical status classification of I-III
3. Single renal stone with a diameter between 2-3 cm confirmed by non-contrast CT scan
4. Signed written informed consent and willingness to comply with study procedures

Exclusion Criteria:

1. Anatomical abnormalities of the urinary tract (e.g., horseshoe kidney, ileal conduit)
2. Uncontrolled urinary tract infection
3. Absolute contraindications for RIRS or PCNL
4. Inability to understand or complete study documentation
5. Failure to follow study protocol or attend follow-up
6. Patients requiring urgent rescue or at high risk for irreversible harm during surgery
7. Patients who voluntarily withdraw from the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Stone-Free Rate (SFR) | 3 months postoperatively
  The proportion of participants who are stone-free after the procedure, defined as no residual stones or residual fragments <2 mm based on postoperative plain abdominal X-ray or non-contrast CT scan.

SECONDARY OUTCOMES:
Incidence of Postoperative Infection (SIRS Criteria) | Within 72 hours postoperatively
  Number and proportion of participants who develop postoperative systemic inflammatory response syndrome (SIRS), defined as meeting at least 2 of the following:
  Temperature >38°C or <36°C
  Heart rate >90 bpm
  Respiratory rate >20/min or PaCO2 <32 mmHg
  WBC count >12×10⁹/L or <4×10⁹/L

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Naval Medical University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skolarikos A, Jung H, Neisius A, et al. EAU Guidelines on Urolithiasis 2024. European Association of Urology. https://uroweb.org/guidelines/urolithiasis
- [Background] Zeng G, Traxer O, Zhong W, Osther P, Pearle MS, Preminger GM, Mazzon G, Seitz C, Geavlete P, Fiori C, Ghani KR, Chew BH, Git KA, Vicentini FC, Papatsoris A, Brehmer M, Martinez JL, Cheng J, Cheng F, Gao X, Gadzhiev N, Pietropaolo A, Proietti S, Ye Z, Sarica K. International Alliance of Urolithiasis guideline on retrograde intrarenal surgery. BJU Int. 2023 Feb;131(2):153-164. doi: 10.1111/bju.15836. Epub 2022 Jul 12. PMID 35733358

DOCUMENTS (1):
  • Study Protocol (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/02/NCT07058402/Prot_000.pdf